CLINICAL TRIAL: NCT06607692
Title: Single-arm Open-label Phase II Study in Children and Adolescents of 177Lu-DOTATATE (Lutathera®) Combined with the PARP Inhibitor Olaparib for the Treatment of Recurrent or Relapsed Solid Tumours Expressing Somatostatin Receptor (SSTR) (LuPARPed)
Brief Title: Study in Children and Adolescents of 177Lu-DOTATATE (Lutathera®) Combined with the PARP Inhibitor Olaparib for the Treatment of Recurrent or Relapsed Solid Tumours Expressing Somatostatin Receptor (SSTR) (LuPARPed).
Acronym: LUPARPED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuPARPed-HM-2024; 2024-512613-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-04; First posted 2024-09-23 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor Cancer; Medulloblastoma; High Risk Neuroblastoma; High Grade Gliomas; Meningioma; Paraganglioma; Pheochromocytoma; Neuroendocrine Tumours (NET); Adrenal Tumours
Keywords: solid tumours; somatostatin receptors; SSTR
MeSH Terms: conditions — Medulloblastoma; Meningioma; Paraganglioma; Pheochromocytoma; Neuroendocrine Tumors; Adrenal Gland Neoplasms | interventions — olaparib; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lu-DOTATATE (Lutathera® ) and olaparib (Experimental): Lu-DOTATATE (Lutathera®) and olaparib for a maximum of 4 cycles unless unacceptable toxic effects occur, there is centrally confirmed disease progression (according to RECIST v1.122) on imaging, the patient is unable or unwilling to adhere to trial procedures, the patient withdraws consent, or the patient dies.
  177Lu-DOTATATE will be administered intravenously, on day 1, every 8 weeks, at a fixed dose of 200 mCi (7.4 GBq) for children >= 12 years old infused intravenously over a period of 30 minutes. For children younger than 12 years old, the dose that will be administered is 200 MBq per kilogram of body weight (maximum 7.4 GBq) infused intravenously over a period of 30 minutes. Concomitant to 177Lu-DOTATATE, patients will receive IV fluids and an IV infusion of amino acid solution for renal protection23. Patients will receive four infusions every 8 weeks (maximum cumulative radioactivity, 29.6 GBq [800 mCi]).
  Olaparib will be administered PO, BID, days 2-29, every 8 weeks
  Interventions: Drug: Olaparib; 177Lu-DOTATATE

INTERVENTIONS:
Drug: Olaparib; 177Lu-DOTATATE — 7Lu-DOTATATE will be administered intravenously, on day 1, every 8 weeks, at a fixed dose of 200 mCi (7.4 GBq) for children >= 12 years old infused intravenously over a period of 30 minutes. For children younger than 12 years old, the dose that will be administered is 200 MBq per kilogram of body weight (maximum 7.4 GBq) infused intravenously over a period of 30 minutes. Concomitant to 177Lu-DOTATATE, patients will receive IV fluids and an IV infusion of amino acid solution for renal protection23. Patients will receive four infusions every 8 weeks (maximum cumulative radioactivity, 29.6 GBq [800 mCi]). Olaparib will be administered PO, BID, days 2-29, every 8 weeks at a fixed dose of 187.5mg/m2 twice daily (BID).

SUMMARY:
Study in children and adolescents of 177Lu DOTATATE (Lutathera®) combined with the PARP inhibitor olaparib for treatment of recurrent or relapsed solid tumours expressing somatostatin receptors (SSTR) (LuPARPed)

DETAILED DESCRIPTION:
Relapsed/refractory (R/R) solid tumours at the paediatric age have a dismal prognosis [5-year overall survival (OS) &lt;20%. There is growing evidence about the somatostatin receptor (SSTR) expression in paediatric tumours, which opens a new diagnostic and therapeutic tool. Somatostatin receptor-targeted therapy with 177Lu-DOTA0-Tyr3-octreotate (177[Lu]Lu DOTA-TATE, 177Lu-DOTATATE, Lutathera®) has been approved by the EMA (2017) and the FDA (2018) for the treatment of adults with midgut neuroendocrine tumours after the excellent results achieved in the phase III NETTER-1 study.

177Lu-DOTATATE is already being explored as monotherapy in children with R/R high-risk neuroblastoma, CNS tumours or meningiomas in 2 pilot studies and 4 clinical trials (ISRCTN98918118, NCT04903899, NCT03966651, NCT05278208). There are two on going clinical trials exploring the recommended phase 2 dose (RP2D) of 177Lu-DOTATATE in children &amp;amp;lt;12 years old, but results are still pending.

The results show promising but insufficient results. Because of its beta particle emission, 177Lu-DOTATATE mainly produces DNA single-strand breaks (SSBs) that are easily repaired by the organism. In order to enhance its effect, the investigators propose its combination with PARP inhibitors (iPARP) so that the SSBs could not be repaired and would lead to the formation of DNA double strand breaks (DSBs) and, subsequently, to cell death. This combination is already being explored in different clinical trials in adults with neuroendocrine tumours and prostate cancer. An interesting study analysed the perfect scheme for the 177Lu-DOTATATE and olaparib combination and concluded that olaparib should be delayed 24 hours after 177Lu-DOTATATE administration in order to facilitate normal tissue repair without decreasing antitumoural activity. It also concludes that there is no benefit in continuing olaparib after 4 weeks of continuous treatment. Olaparib has also been administered in children and there is today a recommended phase 2 dose (187.5 mg/m2 BID)

ELIGIBILITY:
Inclusion Criteria:

* 18 months - 18 years of age at the time of the initial diagnosis.
* ≥ 3 years at the moment of inclusion in the trial.
* Diagnosis: relapsed/refractory solid tumours with positive uptake on SSTR-PET (PET-CT or PET-MRI), performed in the previous three months before entering the study. The positiveness of the study in patients with localized CNS tumours that do not spread through the spine, will be assessed according to:
* Active uptake: when the tumoral lesion shows SSTR expression higher than the one of the background cerebral uptake.
* Negative uptake: when the tumoral lesion shows no SSTR expression. Patients with active uptake in the majority of the tumoral lesions will be considered to have a positive SSTR-PET and will be therefore eligible for the trial.

For the rest of the patients, the evaluation of SSTR expression will be classified according to a qualitative 4-point scale: SSTR expression V (visual score):

* Score = 0: Below or equal to blood pool
* Score = 1: Above blood pool and lower than liver
* Score = 2: Equal to or above liver and lower than spleen
* Score = 3: Equal to or above spleen Patients with scores ≥ 2 in the majority of the tumoral lesions will be considered to have a positive SSTR-PET and will be therefore eligible for the trial. Patients with a higher score are presumed to have a better response to the treatment.
* It is admissible to have non-measurable disease only (e.g., HR-NB with bone-only or bone marrow-only active disease).
* Performance status ≥ 50% according to Lansky scale (<16 years old) or Karnofsky scale (for ≥16 years old).
* Life expectancy of at least 3 months.
* Availability of ability to swallow tablets
* Adequate organ function within 28 days prior to enrolment, as defined by:
* Hb ≥10 g/dl (packed red blood transfusion is acceptable up to 24 hours prior starting treatment);
* White blood cell (WBC) count ≥ 2500/µL (equivalent to 2.5 x 109/L)
* Absolute Neutrophil Count (ANC) ≥ 1000/µl;
* Platelets ≥ 50.000/µl, without transfusion in the prior ≥10 days;
* Serum plasma creatinine ≤ 1.5 x upper limit of normal (ULN) OR estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m2 (assessed by 2009-Schwartz formula).
* Total bilirubin ≤ 1.5 x the institutional ULN. For patients with known Gilbert's Syndrome ≤ 3.0 ULN is permitted.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3.0 ULN OR ≤ 5.0 ULN for patients with liver metastases.
* Albumin >3.0 g/dL (3.0 g/dL is equivalent to 30 g/L)
* A negative serum or urine pregnancy test in women with onset of menses or >12 years of age.
* Patients of reproductive potential must agree to use highly effective contraceptive methods for the entire study duration and up to 7 months, in case of females, and 4 months in case of males, after the last dose of Lutathera, or up to 6 months, in case of females, and 3 months in case of males, after the last dose of olaparib, whichever takes places later.
* Have the ability to comprehend and willingness to provide written informed consent (ICF) for the study before patient registration or any trial-related screening procedures. If the patient is <18 years old, the written informed consent must be signed by the parent(s) or legal guardian(s) according to national regulations. In the case of patients between 12 and 17 years, they must sign an assent form, and if the patient turns 18 during their participation in the study, they must sign an informed consent form.
* Adequate recovery from major surgery prior to receiving study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

* Having received more than one previous treatment with other radiolabelled somatostatin analogues.
* Inability to swallow tablets.
* Subjects who are currently receiving any other anticancer and/or investigational agents. There must be at least two-week of washout from any prior treatment.
* Treatment with long-acting somatostatin analogues within 30 days prior the administration of 177Lu-DOTATATE.
* Known hypersensitivity to any of the excipients.
* Subjects who have an uncontrolled infection.
* Lactating women.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR), measured by RECIST v1.1 | From enrollment up to 12 months after EOT
  The main outcome of the study will be Overall Response Rate (ORR) as measured by RECIST v1.122 . The ORR will be calculated with the corresponding 2-sided 95% Clopper-Pearson exact confidence interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Osuna Marco, PhD, Study Director — HM Monteprincipe
Locations (1):
- HM Monteprincipe, Boadilla del Monte, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided